CLINICAL TRIAL: NCT04001907
Title: Effects of β-hydroxy-β-methyl Butyrate Supplementation and Resistance Exercise on Body Composition, Muscle Strength and Protein Oxidation in Sickle Cell Anaemia.
Brief Title: Effect of Exercise With and Without HMB on Body Composition and Muscle Strength in Sickle Cell Anaemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMB001
Record Dates: First submitted 2019-04-04; First posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-03

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Resistance Training; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise combined with β-hydroxy-β-methylbutyrate (HMB) (Experimental): Resistance Exercise ( 3d/week) and HMB: 3g/d as three 1g capsules orally, for 9 weeks
  Interventions: Behavioral: Resistance exercise; Dietary Supplement: β-hydroxy-β-methylbutyrate
- exercise combined with placebo (Placebo Comparator): Resistance exercise ( 3d/week) and placebo as 3g/d maltodextrin as three 1g capsules orally, for 9 weeks
  Interventions: Behavioral: Resistance exercise; Dietary Supplement: placebo

INTERVENTIONS:
Behavioral: Resistance exercise — effect of exercise and an anabolic agent on body composition, muscle strength, phenylalanine and protein oxidation.
  Other Names: HMB
Dietary Supplement: β-hydroxy-β-methylbutyrate
  Arms: exercise combined with β-hydroxy-β-methylbutyrate (HMB)
Dietary Supplement: placebo
  Other Names: maltodextrin
  Arms: exercise combined with placebo

SUMMARY:
Wasting is a common and significant problem in sickle cell anaemia (SCA) that correlates with poorer clinical outcome such as frequent painful crises, acute chest syndrome and sub normal resistance to infection. Thus, improvement of nutritional status in SCA holds the potential of ameliorating the course of the disease. Elevated haemolysis and its effects are associated with hypermetabolism and have resulted in higher rates of protein breakdown and synthesis, and energy expenditure. Offering more food has not optimized nutritional status and metabolic performance in free-living patients with SCA. Moreover, appetite might be suppressed. Supplementation with β-hydroxy-β-methylbutyrate (HMB), which is produced in the body from leucine, has been shown to have inhibitory effect on protein breakdown and to promote lean tissue synthesis in humans with sarcopenia. Also, HMB has been implicated as an ergogenic tool to promote exercise performance and skeletal muscle hypertrophy. Therefore, the investigators hypothesize that in individuals with SCA, an intervention of resistance exercise with HMB supplement will have a greater enhancing effect on muscle mass and strength compared to receiving resistance exercise without HMB.

DETAILED DESCRIPTION:
The investigators aim to measure muscle strength, body composition and whole body protein oxidation in two groups of adults with SCA within one week before and after 9 weeks of intervention in a randomized, double blinded study. One group (n =12 ) will receive an intervention of resistance exercise and HMB supplement, and the other group (n=12) will receive resistance exercise and a placebo (maltodextrin). Participants will be assigned a study code and all information and samples will be stored under the assigned code.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 18.5 kg/m2

Exclusion Criteria:

* BMI > 19 kg/m2

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-04-30 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Body composition assessment using deuterium dilution method | 3 months
  Change between baseline and after 3 months of intervention
Body composition assessment using Dual-energy X-ray absorptiometry | 3 months
  Change between baseline and after 3 months of intervention
Body composition assessment using bioelectrical impedance | 3 months
  Change between baseline and after 3 months of intervention
muscle strength assessment using the 1-repetition maximum method for the lower body (leg extension and or seated leg press) and upper body (bench press, bicep preacher curl) | 3 months
  Change between baseline and after 3 months of intervention
Protein oxidation using established stable isotope tracer method with oral doses of isotopically labelled sodium bicarbonate and phenylalanine | 3 months
  Change between baseline and after 3 months of intervention

SECONDARY OUTCOMES:
Dietary intake using three 24 h dietary recall before and after intervention | 30 min
  Change between baseline and after 3 months of intervention
Resting metabolic rate using indirect calorimetry before and after intervention | 30 min
  Change between baseline and after 3 months of intervention

OTHER OUTCOMES:
Number of participants with intervention-related abnormal laboratory values as assessed by blood haematology (anaemia profile,white blood cells count, platelet count) | 3 months
  Three measurements at baseline, mid point of intervention and at end of intervention
Number of participants with intervention-related abnormal laboratory values as assessed by blood chemistry (liver function and lipid profile) | 3 months
  Three measurements at baseline, mid point of intervention and at end of intervention
Number of participants with intervention-related adverse effect on emotional profile according to the Circumplex Test of emotion questionnaire | weekly for 3 months
  Assessment at baseline and at the end of each week during the intervention
Number of participants with intervention-related adverse health effect as assessed by completing a health-related questionnaire | weekly for 3 months
  Assessment at baseline and at the end of each week during the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Asha V Badaloo, PhD, Principal Investigator — Tropical Metabolism Research Unit, CAIHR, University of the West Indies; Marvin E Reid, MBBS, PhD, Study Director — Tropical Metabolism Research Unit, CAIHR, University of the West Indies

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson GJ, Wilson JM, Manninen AH. Effects of beta-hydroxy-beta-methylbutyrate (HMB) on exercise performance and body composition across varying levels of age, sex, and training experience: A review. Nutr Metab (Lond). 2008 Jan 3;5:1. doi: 10.1186/1743-7075-5-1. PMID 18173841
- [Background] Badaloo A, Jackson AA, Jahoor F. Whole body protein turnover and resting metabolic rate in homozygous sickle cell disease. Clin Sci (Lond). 1989 Jul;77(1):93-7. doi: 10.1042/cs0770093. PMID 2758764
- [Background] Jackson AA, Landman JP, Stevens MC, Serjeant GR. Urea kinetics in adults with homozygous sickle cell disease. Eur J Clin Nutr. 1988 Jun;42(6):491-6. PMID 3409857
- [Background] Rathmacher JA, Nissen S, Panton L, Clark RH, Eubanks May P, Barber AE, D'Olimpio J, Abumrad NN. Supplementation with a combination of beta-hydroxy-beta-methylbutyrate (HMB), arginine, and glutamine is safe and could improve hematological parameters. JPEN J Parenter Enteral Nutr. 2004 Mar-Apr;28(2):65-75. doi: 10.1177/014860710402800265. PMID 15080599
- [Background] Nissen S, Sharp R, Ray M, Rathmacher JA, Rice D, Fuller JC Jr, Connelly AS, Abumrad N. Effect of leucine metabolite beta-hydroxy-beta-methylbutyrate on muscle metabolism during resistance-exercise training. J Appl Physiol (1985). 1996 Nov;81(5):2095-104. doi: 10.1152/jappl.1996.81.5.2095. PMID 8941534
- [Background] Borack MS, Volpi E. Efficacy and Safety of Leucine Supplementation in the Elderly. J Nutr. 2016 Dec;146(12):2625S-2629S. doi: 10.3945/jn.116.230771. Epub 2016 Nov 9. PMID 27934654
- [Background] Cruz-Jentoft AJ. Beta-Hydroxy-Beta-Methyl Butyrate (HMB): From Experimental Data to Clinical Evidence in Sarcopenia. Curr Protein Pept Sci. 2018;19(7):668-672. doi: 10.2174/1389203718666170529105026. PMID 28554316
- [Background] Heyman MB, Vichinsky E, Katz R, Gaffield B, Hurst D, Castillo R, Chiu D, Kleman K, Ammann AJ, Thaler MM, et al. Growth retardation in sickle-cell disease treated by nutritional support. Lancet. 1985 Apr 20;1(8434):903-6. doi: 10.1016/s0140-6736(85)91677-0. PMID 2858749
- [Background] Di Buono M, Wykes LJ, Ball RO, Pencharz PB. Dietary cysteine reduces the methionine requirement in men. Am J Clin Nutr. 2001 Dec;74(6):761-6. doi: 10.1093/ajcn/74.6.761. PMID 11722957